CLINICAL TRIAL: NCT06124131
Title: Building Engagement Using Financial Incentives Trial - Colorectal Cancer Screening
Acronym: BENEFIT-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2020-1600-BENC; OT2HL158287 (NIH)
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Health Behavior; Colorectal Cancer; Influenza; COVID-19; Vaccine Hesitancy; Vaccine-Preventable Diseases; Healthcare Patient Acceptance
Keywords: Cancer screening; Preventive healthcare; Vaccine uptake; Patient financial incentives; Federally qualified health center; Health services
MeSH Terms: conditions — Health Behavior; Colorectal Neoplasms; Influenza, Human; COVID-19; Vaccination Hesitancy; Vaccine-Preventable Diseases; Patient Acceptance of Health Care | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to a study arm for the duration of their two months in the study
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Primary care outreach staff will recruit and randomize participants and deliver the intervention. Group assignment will be documented in a separate study database not accessible by the primary care provider. Outcomes will be assessed in electronic health records data, which will be queried by primary care staff who do not have access to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full financial incentives (Experimental): $50/service patient financial incentive for completion of: COVID-19 shot, flu shot, colorectal cancer screening
  Interventions: Behavioral: Financial incentive for colorectal cancer screening; Behavioral: Financial incentive for flu shot; Behavioral: Financial incentive for COVID-19 shot
- Partial financial incentives (Active Comparator): $50/service patient financial incentive for completion of: COVID-19 shot, flu shot
  Interventions: Behavioral: Financial incentive for flu shot; Behavioral: Financial incentive for COVID-19 shot

INTERVENTIONS:
Behavioral: Financial incentive for colorectal cancer screening — $50 incentive paid to participant for completion of colorectal cancer screening within 2 months of enrollment
  Arms: Full financial incentives
Behavioral: Financial incentive for flu shot — $50 incentive paid to participant for completion of flu shot within 2 months of enrollment
Behavioral: Financial incentive for COVID-19 shot — $50 incentive paid to participant for completion of COVID-19 shot within 2 months of enrollment

SUMMARY:
The goal of this pilot clinical trial is to determine feasibility and explore whether financial incentives paid to primary care patients for completing colorectal cancer screening increase completion of colorectal cancer screening. The main questions it aims to answer are:

* Do patient financial incentives for completing colorectal cancer screening increase screening completion?
* Does a patient financial incentive for colorectal cancer screening offered alongside patient financial incentives for COVID-19 and flu shots increase completion of those shots?

Participants who are due for colorectal cancer screening will receive telephone outreach from primary care staff who will offer a stool-based colorectal cancer screening. Participants will be randomly assigned to either Group 1 or Group 2. Group 1 participants will be offered financial incentives for completing COVID-19 and flu shots within 2 months of enrollment. Group 2 participants will be offered financial incentives for completing a COVID-19 shot, a flu shot, and colorectal cancer screening within 2 months of enrollment.

Researchers will compare to see if completion of a COVID-19 shot, a flu shot, and colorectal cancer screening is different between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 to 75
* Receive care at participating primary care clinic
* Due for colorectal cancer screening
* Ability to understand and speak English

Exclusion Criteria:

* Currently participating in another clinical trial or research study on colorectal cancer screening
* Unable or unwilling to give informed consent

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie A Krousel-Wood, MD, MSPH, Principal Investigator — Tulane University
Locations (1):
- Tulane University School of Medicine, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Full Financial Incentives | Partial Financial Incentives
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Financial Incentives | Partial Financial Incentives | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.48 (6.63) | 52.32 (6.74) | 52.40 (6.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 35
  Male | 10 | 5 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 11 | 21
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 24 | 25 | 49
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Difference in Percent of Participants Completing Colorectal Cancer Screening Between Study Arms
Description: Completion of colonoscopy, sigmoidoscopy, CT colonography, or stool-based colorectal cancer screening test as documented in electronic health record within two months of study enrollment
Time Frame: Two months
Measure: Count of Participants; unit: Participants
Arm/Group | Full Financial Incentives | Partial Financial Incentives
Number analyzed (Participants) | 25 | 25
Participants | 17 | 8

2. Secondary Outcome: Difference in Percent of Participants Completing COVID-19 Shot Between Study Arms
Description: Completion of COVID-19 shot as documented in electronic health record within two months of study enrollment
Time Frame: Two months
Measure: Count of Participants; unit: Participants
Arm/Group | Full Financial Incentives | Partial Financial Incentives
Number analyzed (Participants) | 25 | 25
Participants | 1 | 0

3. Secondary Outcome: Difference in Percent of Participants Completing Flu Shot Between Study Arms
Description: Completion of flu shot as documented in electronic health record within two months of study enrollment
Time Frame: Two months
Measure: Count of Participants; unit: Participants
Arm/Group | Full Financial Incentives | Partial Financial Incentives
Number analyzed (Participants) | 25 | 25
Participants | 9 | 10

4. Secondary Outcome: Difference in Percent of Participants Completing at Least One of the Following Services Between Study Arms: Colorectal Cancer Screening, COVID-19 Shot, Flu Shot
Description: Completion of colorectal cancer screening (colonoscopy, sigmoidoscopy, CT colonography, or stool-based colorectal cancer screening test), COVID-19 shot, *OR* flu shot as documented in electronic health record within two months of study enrollment
Time Frame: Two months
Measure: Count of Participants; unit: Participants
Arm/Group | Full Financial Incentives | Partial Financial Incentives
Number analyzed (Participants) | 25 | 25
Participants | 20 | 13

5. Secondary Outcome: Difference in Percent of Participants Completing All Three Services Between Study Arms: Colorectal Cancer Screening, COVID-19 Shot, Flu Shot
Description: Completion of colorectal cancer screening (colonoscopy, sigmoidoscopy, CT colonography, or stool-based colorectal cancer screening test), COVID-19 shot, *AND* flu shot as documented in electronic health record within two months of study enrollment
Time Frame: Two months
Measure: Count of Participants; unit: Participants
Arm/Group | Full Financial Incentives | Partial Financial Incentives
Number analyzed (Participants) | 25 | 25
Participants | 1 | 0

6. Other Pre Specified Outcome: Number of Patients Reached for Recruitment
Description: Number of patients reached for recruitment
Time Frame: Three months
Population: Overall Number of Participants Analyzed represents all patients who were approached and considered for recruitment.
Measure: Count of Participants; unit: Participants
Groups:
- Recruitment Sample: Patients approached
Arm/Group | Recruitment Sample
Number analyzed (Participants) | 123
Participants | 107

7. Other Pre Specified Outcome: Number of Patients Assessed for Eligibility
Description: Number of patients assessed for eligibility
Time Frame: Three months
Population: Overall Number of Participants Analyzed represents all patients who were reached during recruitment
Measure: Count of Participants; unit: Participants
Groups:
- Reachable Sample: Patients who were reached
Arm/Group | Reachable Sample
Number analyzed (Participants) | 107
Participants | 93

8. Other Pre Specified Outcome: Number of Patients Consented and Randomized
Description: Number of patients consented and randomized
Time Frame: Three months
Population: Overall Number of Participants Analyzed represents all patients who underwent eligibility screening and were eligible to participate.
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Sample: Patients who underwent eligibility screening were eligible to participate.
Arm/Group | Eligible Sample
Number analyzed (Participants) | 53
Participants | 50

9. Other Pre Specified Outcome: Number of Patients Who Receive the Outreach Call Intervention
Description: Number of patients who receive the outreach call intervention
Time Frame: Three months
Measure: Count of Participants; unit: Participants
Arm/Group | Full Financial Incentives | Partial Financial Incentives
Number analyzed (Participants) | 25 | 25
Participants | 25 | 25

ADVERSE EVENTS:
Time Frame: Two months
Description: All-Cause Mortality was assessed/monitored using the primary care clinic electronic health record (EHR). Serious and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Full Financial Incentives | Partial Financial Incentives
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT06124131/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT06124131/SAP_001.pdf